CLINICAL TRIAL: NCT00004276
Title: Phase II Placebo Controlled Study of Thalidomide in Patients With Mycobacterial and HIV Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Rockefeller University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11682; RU-0300395
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: HIV Infections; Mycobacterium Infections; Tuberculosis
Keywords: bacterial infection; human immunodeficiency virus infection; immunologic disorders and infectious disorders; mycobacterium infection; mycobacterium tuberculosis infection; rare disease; viral infection
MeSH Terms: conditions — HIV Infections; Mycobacterium Infections; Tuberculosis; Bacterial Infections; Acquired Immunodeficiency Syndrome; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
OBJECTIVES: I. Evaluate whether thalidomide modulates toxic host inflammatory responses in patients receiving antitubercular therapy.

II. Evaluate whether thalidomide modifies tumor necrosis factor-mediated toxic symptoms of HIV and mycobacterial infections, and limits progression of HIV immunodeficiency.

III. Evaluate whether thalidomide stimulates immunity in patients with HIV and/or mycobacterial infections.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind study. Patients are stratified by type of infection.

Patients are randomly assigned to oral thalidomide or placebo. Therapy is administered daily for up to 8 weeks, beginning the night before antitubercular treatment is initiated.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Human immunodeficiency virus (HIV) or mycobacterial infection that requires at least 10 days of inpatient antitubercular treatment

Mycobacterial infection confirmed by positive acid-fast bacilli smear or culture for Mycobacterium tuberculosis

At least 1 of the following signs and symptoms required:

* Temperature over 38 degrees C on at least 2 occasions within 1 week prior to treatment
* Weight loss greater than 5 kg
* Pulmonary involvement in at least 1 lobe on x-ray

Night sweats on at least 2 occasions within 1 week prior to treatment

--Prior/Concurrent Therapy--

Concurrent rifampicin, isoniazid, pyrazinamide, and ethambutol for tuberculosis allowed

--Patient Characteristics--

* No neuropathy and not at risk for neuropathy
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1990-09; Study Completion 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Gilla Kaplan, Study Chair — Rockefeller University

REFERENCES:
- [Background] Haslett P, Tramontana J, Burroughs M, Hempstead M, Kaplan G. Adverse reactions to thalidomide in patients infected with human immunodeficiency virus. Clin Infect Dis. 1997 Jun;24(6):1223-7. doi: 10.1086/513665. PMID 9195087
- [Background] Tramontana JM, Utaipat U, Molloy A, Akarasewi P, Burroughs M, Makonkawkeyoon S, Johnson B, Klausner JD, Rom W, Kaplan G. Thalidomide treatment reduces tumor necrosis factor alpha production and enhances weight gain in patients with pulmonary tuberculosis. Mol Med. 1995 May;1(4):384-97. PMID 8521296
- [Background] Haslett P, Hempstead M, Seidman C, Diakun J, Vasquez D, Freedman VH, Kaplan G. The metabolic and immunologic effects of short-term thalidomide treatment of patients infected with the human immunodeficiency virus. AIDS Res Hum Retroviruses. 1997 Aug 10;13(12):1047-54. doi: 10.1089/aid.1997.13.1047. PMID 9264292
- [Background] Bekker LG, Haslett P, Maartens G, Steyn L, Kaplan G. Thalidomide-induced antigen-specific immune stimulation in patients with human immunodeficiency virus type 1 and tuberculosis. J Infect Dis. 2000 Mar;181(3):954-65. doi: 10.1086/315328. PMID 10720518
- [Background] Klausner JD, Makonkawkeyoon S, Akarasewi P, Nakata K, Kasinrerk W, Corral L, Dewar RL, Lane HC, Freedman VH, Kaplan G. The effect of thalidomide on the pathogenesis of human immunodeficiency virus type 1 and M. tuberculosis infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Mar 1;11(3):247-57. doi: 10.1097/00042560-199603010-00005. PMID 8603261